CLINICAL TRIAL: NCT00229931
Title: The Role of Triamcinolone Injection During Cataract Extraction for Diabetic Patients With Pre-Operative Macular Edema
Brief Title: Triamcinolone vs. Laser for Diabetic Macular Edema
Acronym: IVTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2746
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: DIABETIC MACULAR EDEMA
Keywords: CATARACT EXTRACTION; MACULAR EDEMA; DIABETES; FOCAL LASER; TRIAMCINOLONE
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus | interventions — Triamcinolone Acetonide; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser therapy (Active Comparator): If randomized to laser therapy at time of cataract surgery, laser therapy will be performed one month after cataract surgery. If macular edema does not respond an additional laser therapy will be performed. If macular edema persists after 2 lasers, then IVTA will be administered as per standard of care.
  Interventions: Procedure: laser
- Triamcinolone therapy (Active Comparator): At time of cataract surgery, will have IVTA injection. If macular edema does not show improvement at 1 month, then can have repeat IVTA injection. If the macular edema is stil not improved after 2nd injection, participant will be considered "treatment failure" and will be given the option to have laser therapy.
  Interventions: Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: Triamcinolone acetonide — 4mg of intravitreal triamcinolone at time of cataract surgery with option to repeat at one month if no response
  Other Names: Kenalog
  Arms: Triamcinolone therapy
Procedure: laser — Laser treatment 1 month after cataract surgery with option to repeat once if no improvement.
  Other Names: focal laser photocoagulation
  Arms: Laser therapy

SUMMARY:
The purpose of this study is to determine if intravitreal triamcinolone acetonide (IVTA) injection at the time of cataract surgery will improve visual acuity and decrease post-operative swelling in diabetic patients requiring cataract extraction as compared to the conventional treatment of laser following cataract surgery.

The subjects will be followed for 11 visits over 3 year. Visits will occur at screening,1, 3,6,9,12,18,24,30 and 36 months post surgery.

DETAILED DESCRIPTION:
Protocol Summary:

This is a randomized, prospective study comparing diabetic patients with pre-operative macular edema undergoing cataract surgery treated with either 4 mg of intravitreal triamcinolone at the time of cataract surgery or focal laser treatment 1 month following cataract surgery.

Disease State:

The conventional treatment for clinically significant macular edema is focal laser photocoagulation. In some diabetic patients however, the cataract often impedes fundus visualization for optimal laser treatment. In these patients focal laser treatment is deferred until after cataract surgery.

Study aim:

The purpose of this study is to determine if intravitreal triamcinolone acetonide (IVTA) injection at the time of cataract surgery will improve visual acuity and decrease post-operative macular edema in diabetic patients with pre-operative macular edema requiring cataract extraction as compared to the conventional treatment of focal laser photocoagulation following cataract surgery.

Hypothesis:

We propose that by injecting triamcinolone intravitreally at the time of cataract surgery in patients who have pre-operative macular edema, we will not only reduce the risk of exacerbating macular edema but also possibly improve the final visual outcome.

Study Procedures:

After informed consent is obtained each patient will be placed, based on a randomization scheme, into either the control group receiving the conventional focal laser treatment one month following cataract extraction or into the study group receiving the IVTA injection at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* visually significant cataracts
* pre-operative visual acuity 20/50 or worse
* pre-operative optical coherence tomography (OCT) showing at least 250 microns central foveal thickness.

Exclusion Criteria:

* macular ischemia
* vitreomacular traction
* macular hole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Leonard, MD, Principal Investigator — Dean A. McGee Eye Institute
Locations (1):
- Dean A. McGee Eye Institute, Oklahoma City, Oklahoma, United States

REFERENCES:
- See also: Dean McGee Eye Institute — http://www.dmei.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser Therapy | Triamcinolone Therapy
Started | 6 | 5
Completed | 2 | 3
Not Completed | 4 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser Therapy | Triamcinolone Therapy | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Main Outcome Measures Will be Quantitative Changes in OCT Central Thickness, Visual Acuity, and Number of Snellen Acuity Lines Gained/Lost.
Time Frame: 3 years
Population: Due to lack of follow up from patients, this outcome was not analyzed; data were not collected
Arm/Group | Laser Therapy | Triamcinolone Therapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Rate of Elevated Intraocular Pressures, Retinal Detachment, Infection, and Vitreous Hemorrhage.
Time Frame: 3 years
Population: Data were not collected
Arm/Group | Laser Therapy | Triamcinolone Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Laser Therapy | Triamcinolone Therapy
All-Cause Mortality (participants affected / at risk) | 2/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser Therapy (N=6) | Triamcinolone Therapy (N=5)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for shortness of breath
Kidney Failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for kidney failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser Therapy (N=6) | Triamcinolone Therapy (N=5)
Vitreous Hemorrhage (Eye disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to lack of patient follow up on this study, sufficient data was not available for analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No